CLINICAL TRIAL: NCT04852783
Title: US IDE Study of the Contour NEurovasCular System™ for IntraCranial Aneurysm Repair
Acronym: NECC
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cerus Endovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNX102-01
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aneurysm, Intracranial
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, multicenter single-arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Attempted to Treat (Experimental): Attempted to treat (ATT) with the investigational device
  Interventions: Device: Contour Neurovascular System

INTERVENTIONS:
Device: Contour Neurovascular System — Endovascular embolization of wide-necked, bifurcated saccular intracranial aneurysms.

SUMMARY:
The purpose of this trial is to gather data on the safety and effectiveness of the Contour /Contour 021 System in the treatment of wide-necked bifurcated saccular, intracranial aneurysms for submission to FDA in support of a premarket approval application for the device.

DETAILED DESCRIPTION:
The purpose of this trial is to gather data on the safety and effectiveness of the Contour /Contour 021 System in the treatment of wide-necked bifurcated saccular, intracranial aneurysms for submission to FDA in support of a premarket approval application for the device. This trial is a prospective, multicenter single-arm study. Up to 220 subjects will be enrolled at up to 20 participating investigational sites.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18-75 years of age at the time of screening.
2. Patient has a single ruptured or unruptured IA requiring treatment. If the patient has an additional IA requiring treatment, the additional IA must not require treatment within 60 days of the index procedure.
3. The target IA must have the following characteristics:

   * Saccular morphology
   * Located at a bifurcation in the anterior or posterior circulation
   * Aneurysm neck diameter between 2 and 10 mm and aneurysm equatorial diameter between 2 and 10.5 mm
   * Wide-necked, defined as neck size ≥ 4 mm or a dome/neck ratio < 2
4. Patient may be treated with Contour without the use of additional implanted devices.
5. Patient is able to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule.
6. Patient or legally authorized representative has signed and dated an institutional review board (IRB)/Ethics Committee (EC)-approved written informed consent prior to initiation of any study procedures.

   FOR PATIENTS WITH UNRUPTURED ANEURYSM
7. Patient meets the criteria outlined in the "Guidelines for the Management of Patients With Unruptured Intracranial Aneurysms" as published by the AHA/ASA FOR PATIENTS WITH RUPTURED ANEURYSM
8. Patient meets the criteria outlined in the "Guidelines for the Management of Aneurysmal Subarachnoid Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association" as published by the AHA/ASA.
9. Patient must be neurologically stable with Hunt & Hess Score of I, II or III.

Exclusion Criteria:

1. Anatomy or physiology considered unsuitable for endovascular treatment with the Contour device by the implanting physician and/or the Patient Selection Committee
2. Target IA contains other devices/implants (e.g., coils) that could interfere with the correct placement of the Contour device
3. Subject has a known, untreatable hypersensitivity to contrast dye, iodine, or any component of the treatment device.
4. Contraindication to anticoagulants or anti-platelet medications
5. Stenosis of the target IA's parent vessel is >50%
6. Anticoagulation medications (e.g., warfarin) that cannot be discontinued
7. Acute / chronic renal failure (unless on dialysis) and/or creatinine > 2.00 mg/dl or > 182 μmol/L
8. Vascular disease or other vascular anomaly that precluded the necessary access to the aneurysm for use of the study device.
9. Clinical, angiographic or CT evidence of vasospasm, vasculitis, an intracranial tumor (except small meningioma) or any other intracranial vascular malformations on presentation.
10. Conditions placing them at high risk for ischemic stroke or had exhibited ischemic symptoms such as transient ischemic attacks, minor strokes, or stroke-in-evolution within the prior 60-days.
11. Any circulatory, neurovascular, cardiovascular, or neurologic conditions that can result in unstable neurological symptoms (e.g., multiple sclerosis, established seizure disorder).
12. modified Rankin Scale (mRS) score ≥ 2 prior to presentation or rupture (as applicable).
13. SAH from a non-index aneurysm or any other intracranial hemorrhage within 90 days.
14. Physical, neurologic or psychiatric conditions which precluded his/her ability to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule.
15. Pregnant, breastfeeding or planning pregnancy in the next 2 years
16. Subject is enrolled in another device or drug study in which participation could confound study results.
17. Life expectancy of less than 2 years due to an illness or condition other than the index intracranial aneurysm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Death or stroke within 30 days of treatment or ipsilateral stroke or neurological death between 30 days and 1 year. | 30 days
  Death or stroke within 30 days of treatment or ipsilateral stroke or neurological death between 30 days and 1 year.
Primary Effectiveness Endpoint: Complete occlusion of the aneurysm with Contour without retreatment, recurrent subarachnoid hemorrhage, or significant parent artery stenosis at one (1) year after treatment as assessed by the angiographic core laboratory. | 1 year
  Complete occlusion of the aneurysm with Contour as defined by complete aneurysm occlusion (Raymond Roy Scale , of 1) without retreatment, recurrent subarachnoid hemorrhage, or significant parent artery stenosis (> 50% stenosis) at one (1) year after treatment as assessed by the angiographic core laboratory.

SECONDARY OUTCOMES:
Key Secondary Effectiveness Endpoint | 1 year
  The trial's secondary endpoint is the proportion of subjects with angiographic aneurysmal recurrence defined as aneurysm growth or recanalization at one (1) year after treatment.
Key Secondary Safety Endpoint | 1 year
  Proportion of subjects with death of any non-accidental cause or any major stroke (an ischemic or hemorrhagic stroke resulting in an increase of 4 points or more on the NIHSS as of day 7 post onset) within the first 30-days after treatment or major ipsilateral stroke or death due to neurologic cause from day 31 to 365 after treatment.
  A major stroke is "a stroke, which increased the NIHSS by ≥ 4 at the time of assessment and which remained present after 7 days"

CONTACTS AND LOCATIONS:
Overall Officials: Pascal M Jabbour, MD, Principal Investigator — Jefferson University Hospitals; Demetrius Lopes, MD, Principal Investigator — Advocate Medical Group - Brain and Spine Institute
Locations (20):
- United States (20):
  - Swedish Medical Center, Englewood, Colorado
  - Baptist Health, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Advocate Aurora Health, Park Ridge, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMASS Medical Center, Worcester, Massachusetts
  - University at Buffalo Neurosurgery, Buffalo, New York
  - NYU Langone Health, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - NC Heart and Vascular Research LLC, Raleigh, North Carolina
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Alejandro Spiotta, Charelston, South Carolina
  - Semmes-Murphy Clinic, Memphis, Tennessee
  - Medical City Plano, Plano, Texas
  - Swedish Neuroscience Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No